CLINICAL TRIAL: NCT05902546
Title: Effect of High Intensity Interval Training Versus Moderate Intensity Aerobic Exercise on Insulin Resistance in Type 2 Diabetes
Brief Title: Effect of HIIT Vs Moderate Intensity Aerobic Exercise on Insulin Resistance in Type 2 DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Collaborators: Ahmed Maher Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Mina Atef Georgui Elias, Lecturer Internal Medicine & Geriatrics, Faculty of Physical Therapy, Badr University in Cairo., Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-230507-21
Record Dates: First submitted 2023-06-03; First posted 2023-06-15 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (group A) (Experimental): 30 Diabetic patients (Type 2 Diabetes Mellitus) will receive high intensity interval training
  Interventions: Other: High intensity interval training
- moderate intensity aerobic exercise (group B) (Experimental): 30 Diabetic patients (Type 2 Diabetes Mellitus) will receive moderate intensity aerobic exercise
  Interventions: Other: moderate intensity aerobic exercise

INTERVENTIONS:
Other: High intensity interval training — Patients will receive interval training exercise of high intensity. This includes several rounds that alternate between several minutes of high intensity movements to significantly increase the heart rate to at least 80% of one's maximum heart rate, followed by short periods of rest
  Arms: High intensity interval training (group A)
Other: moderate intensity aerobic exercise — Patients will receive moderate intensity continuous aerobic exercise (walking) for 40 minutes (preceded by 10 minutes warming up and followed by 5 minutes cooling down)
  Arms: moderate intensity aerobic exercise (group B)

SUMMARY:
Comparing between the efficacy of high intensity interval training and moderate intensity aerobic exercises on insulin resistance in type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The study aims at differentiating between high intensity interval training and moderate intensity continuous aerobic exercise in terms of their effect of Insulin resistance in patients diagnosed with type 2 Diabetes Mellitus. All participants will have lab analysis for Serum Homa-IR prior to intervention and after 1 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus Patients.
* Diagnosed for more than 1 years at the time of the study.
* Patients with fair control of blood glucose using hypoglycemic drugs

Exclusion Criteria:

* Type 1 (Insulin Dependant) Diabetes Mellitus patients.
* Patients with disability that can't perform exercises.
* Patient with known Cardiovascular diseases.
* Patients with kidney/liver diseases

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance (Homa-IR) | 1 month
  Serum insulin resistance indicator (Homa-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Mina AG Elias, Dr., Principal Investigator — Dept of Internal Medicine & geriatric, Faculty of Physical Therapy, Badr University in Cairo, Egypt.; Khaled M Mounir, Dr., Study Chair — Dept of Cardiopulmonary & internal medicine rehab, Faculty of Physical Therapy, Galala Univ; Egypt.
Locations (4):
- Egypt (4):
  - Ahmed Maher Teaching Hospital, Cairo
  - Elamahaba Specialized Charity Polyclinics, Cairo
  - Trust Physical Therapy Center and Rehabilitation, Cairo
  - Badr University in Cairo, Faculty of Physical Therapy, Outpatient Clinic, Cairo

IPD SHARING:
Plan to Share IPD: No